CLINICAL TRIAL: NCT03848182
Title: Analysis of T Cells to Tetanus Toxoid Antigens in Patients With Pancreatic Cancer Treated With Gemcitabine
Brief Title: Analyzing Childhood Recall Antigens in Patients With Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Pancreatic Cancer Action Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016-7197; 422247 (Other Grant/Funding Number: Pancreatic Cancer Action Network)
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer
Keywords: T-cell responses; Pancreatic cancer; Gemcitabine; Perforin; Granzyme-B; Myeloid-derived suppressor cells
MeSH Terms: conditions — Pancreatic Neoplasms; Lipodystrophy, Congenital Generalized | interventions — Gemcitabine; Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Gemcitabine with TT vaccine booster (Experimental): Gemcitabine will be delivered as is standard of care. Patients diagnosed with pancreatic ductal carcinoma (PCD) will be treated with Gemcitabine and boosted once with the human childhood vaccine to TT
  Interventions: Drug: Gemcitabine; Biological: TT vaccine booster

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine will be administered on days 1, 8, 15 every 28 days
  Other Names: Gemzar
Biological: TT vaccine booster — One human TT childhood vaccine booster will be administered on day 8
  Other Names: Tetanus vaccine

SUMMARY:
The investigator is developing an immune therapy against pancreatic cancer. Immune cells, known as "T cells with tumor killing capacity", are involved in this immune therapy. In mice with pancreatic cance there is evidence that one tetanus toxoid (TT) vaccination (that patients receive from childhood) combined with Gemcitabine activates these killer T cells. (Gemcitabine improves T cell responses) These killer T cells are able to destroy tumor cells uploaded with TT protein (such studies are planned in future clinical trials). The goal of this study is to test whether one TT vaccination combined with Gemcitabine treatment activates the same T cells in pancreatic cancer patients.

DETAILED DESCRIPTION:
Treating PDAC patients with gemcitabine and one TT booster Gemcitabine will be delivered as is standard of care. However, doses may be modified by the treating physician based on patient tolerance. Patients diagnosed with PDAC will be treated with Gemcitabine and boosted once with the human childhood vaccine to TT by Dr. Chuy as outlined in Fig 2. Gemcitabine will be administered on days 1, 8, 15 every 28 days, and one booster with the human TT childhood vaccine will be administered on day 8 (there must be 2 hrs between the TT booster and the Gemcitabine treatment). Blood will be drawn just before each Gemcitabine treatment, except on day 8 at least 2 hrs will be needed between the blood draw and Gemcitabine treatment because the TT booster needs to be given just after the blood draw but 2 hrs before the Gemcitabine treatment (Fig 2). Three tubes of 10 mls each with heparinized blood will be needed for the isolation of peripheral blood mononuclear cells (PBMC). Two tubes will be used to analyze the T cells and one tube for analyzing the MDSC. The memory T cells and MDSC will be analyzed in the laboratory of Dr. Gravekamp.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the pancreas
2. Patients is a candidate for gemcitabine chemotherapy (adjuvant, metastatic, locally advanced, borderline resectable settings all permitted)
3. Patients at least 18 years of age
4. ECOG performance status 0-2
5. Consent to donate 12 tubes of peripheral blood of 10 mL each
6. Adequate organ function as defined as -neutrophil count ≥ 1200 -platelets ≥ 75,000 -hemoglobin ≥ 8.0 -bilirubin ≤ 2.0 -creatinine ≤2.0 or calculated GFR ≥ 30
7. Ability to understand and willingness to sign a written informed consent document
8. Prior chemotherapy permitted, as long as 60 days have lapsed since last dose. Prior radiation therapy permitted, as long as 28 days lapsed since last treatment.
9. Patients may receive other concurrent chemotherapy, immunotherapy, or radiotherapy

Exclusion Criteria:

1. Patients never been immunized with tetanus toxoid (TT). Patients with a history of adverse reaction to tetanus vaccine (with the exception of self-limited fever or local tissue reaction
2. Patients may not be receiving any investigational agents
3. Pregnant women
4. Patients with HIV

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Gravekamp, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients diagnosed with PDAC will be treated with Gemcitabine as is standard of care on days 1, 8, 15 every 28 days. On day 8 one booster with the human TT childhood vaccine will be administered.
  Blood will be drawn before each Gemcitabine treatment. On day 8, TT booster will be administered immediately after blood draw but at least 2 hours before Gemcitabine treatment. Patients who withdraw on or before Day 8 (before TT treatment) will not be included in data analysis.
Period: Overall Study
Arm/Group | Gemcitabine With TT Vaccine Booster
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Patients are evaluated as is standard of care for patients receiving gemcitabine chemotherapy
Arm/Group | Gemcitabine With TT Vaccine Booster
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 2
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in CD4 T Cell Responses Before TT Booster
Description: The relative difference in CD4 T cell counts before and after administration of the TT booster vaccine (Day 8) will be compared. The number of cells per microliter (cells/µL) will be determined. The proportion of at least 3-fold increase will be reported along with its 95% CI. The actual magnitude of change will be examined by taking a log scale of CD4 counts and report a mean of change on CD4 on its log scale along with its 95% CI.
Time Frame: Day 1
Population: Blood samples were collected and analyzed from 10 patients by flow cytometry as well as by ELISPOT.
Measure: Mean (Standard Deviation); unit: cells/uL
Groups:
- Gemcitabine With TT Vaccine Booster: Gemcitabine will be delivered as is standard of care. Patients diagnosed with pancreatic ductal carcinoma (PCD) will be treated with Gemcitabine and boosted once with the human childhood vaccine to TT
  Gemcitabine: Gemcitabine will be administered on days 1, 8, 15 and every 28 days
  TT vaccine booster: One human TT childhood vaccine booster will be administered on day 8
Arm/Group | Gemcitabine With TT Vaccine Booster
Number analyzed (Participants) | 10
cells/uL | NA (NA) — Due to the condition of the blood samples analytical results were unable to be interpreted. As such, data is not available and mean CD4 T cell results have been identified as 'NA'.

2. Primary Outcome: Change in CD4 T Cell Responses Before TT Booster
Description: as for outcome 1
Time Frame: Day 8
Population: Blood samples were collected and analyzed by flow cytometry as well as by ELISPOT.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Gemcitabine With TT Vaccine Booster
Number analyzed (Participants) | 10
cells/uL | NA (NA) — Due to the condition of the blood samples analytical results were unable to be interpreted. As such, data is not available and mean CD4 T cell results have been identified as 'NA'.

3. Primary Outcome: Change in CD4 T Cell Responses After TT Booster
Description: as for outcome 1
Time Frame: Day 15
Population: Blood samples were collected and analyzed by flow cytometry as well as by ELISPOT.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Gemcitabine With TT Vaccine Booster
Number analyzed (Participants) | 10
cells/uL | NA (NA) — Due to the condition of the blood samples analytical results were unable to be interpreted. As such, data is not available and mean CD4 T cell results have been identified as 'NA'.

4. Primary Outcome: Change in CD4 T Cell Responses After TT Booster
Description: as for outcome 1
Time Frame: Day 28
Population: Blood samples were collected and analyzed by flow cytometry as well as by ELISPOT.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Gemcitabine With TT Vaccine Booster
Number analyzed (Participants) | 10
cells/uL | NA (NA) — Due to the condition of the blood samples analytical results were unable to be interpreted. As such, data is not available and mean CD4 T cell results have been identified as 'NA'.

5. Secondary Outcome: Change in CD8 T Cell Responses Before TT Booster
Description: The relative difference in CD8 T cell counts before and after administration of the TT booster vaccine (Day 8) will be compared. The number of cells per microliter (cells/µL) will be determined. The proportion of at least 3-fold increase will be reported along with its 95% CI. The actual magnitude of change will be examined by taking a log scale of CD8 counts and report a mean of change on CD8 on its log scale along with its 95% CI.
Time Frame: Day 1
Population: Blood samples were collected and analyzed by flow cytometry as well as by ELISPOT.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Gemcitabine With TT Vaccine Booster
Number analyzed (Participants) | 10
cells/uL | NA (NA) — Due to the condition of the blood samples analytical results were unable to be interpreted. As such, data is not available and mean CD4 T cell results have been identified as 'NA'.

6. Secondary Outcome: Change in CD8 T Cell Responses Before TT Booster Vaccine
Description: as for outcome 5
Time Frame: Day 8
Population: Blood samples were collected and analyzed by flow cytometry as well as by ELISPOT.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Gemcitabine With TT Vaccine Booster
Number analyzed (Participants) | 10
cells/uL | NA (NA) — Due to the condition of the blood samples analytical results were unable to be interpreted. As such, data is not available and mean CD4 T cell results have been identified as 'NA'.

7. Secondary Outcome: Change in CD8 T Cell Responses After TT Booster
Description: as for outcome 5
Time Frame: Day 15
Population: Blood samples were collected and analyzed by flow cytometry as well as by ELISPOT.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Gemcitabine With TT Vaccine Booster
Number analyzed (Participants) | 10
cells/uL | NA (NA) — Due to the condition of the blood samples analytical results were unable to be interpreted. As such, data is not available and mean CD4 T cell results have been identified as 'NA'.

8. Secondary Outcome: Change in CD8 T Cell Responses After TT Booster
Description: as for outcome 5
Time Frame: Day 28
Population: Blood samples were collected and analyzed by flow cytometry as well as by ELISPOT.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Gemcitabine With TT Vaccine Booster
Number analyzed (Participants) | 10
cells/uL | NA (NA) — Due to the condition of the blood samples analytical results were unable to be interpreted. As such, data is not available and mean CD4 T cell results have been identified as 'NA'.

9. Other Pre Specified Outcome: Change in Myeloid-derived Suppressor Cells
Time Frame: Day 8
Population: MDSC data was not collected or analyzed for this study.
Arm/Group | Gemcitabine With TT Vaccine Booster
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 month following Gemcitabine administration, for a total of up to 2 months
Description: Adverse events were reported and coded using the Modified NCI Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Version 4.0
Arm/Group | Gemcitabine With TT Vaccine Booster
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine With TT Vaccine Booster (N=10)
Gallbladder Perforation (Hepatobiliary disorders) | 1 (1) — Verbatim Term: Perforated Gall Bladder
Duodenal Hemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine With TT Vaccine Booster (N=10)
Fatigue (General disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 8 — Verbatim Terms: Abdominal Pain, Intermittent Abdominal Pain, Abdominal Discomfort
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 — Verbatim Terms: Dyspnea, Shortness of Breath
Chest Pain (Cardiac disorders) | 2 — Verbatim Terms: Chest Pain, Occasional Chest Pain
Constipation (Gastrointestinal disorders) | 3
Edema Limbs (General disorders) | 1 — Verbatim Term: Bilateral Lower Extremity Edema
Anorexia (Metabolism and nutrition disorders) | 3
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 5 — Verbatim Term: Weakness
Cough (Respiratory, thoracic and mediastinal disorders) | 2 — Verbatim Terms: Intermittent Cough, Blood-tinged Cough
Poor Appetite (Metabolism and nutrition disorders) | 5 — Verbatim Terms: Poor Appetite, Poor PO Intake, Appetite Change
Weight Loss (Investigations) | 4 — Verbatim Terms: Weight Loss, Weight Loss (>40lbs in one month)
Gait Disturbance (General disorders) | 3 — Verbatim Term: Gait Problem
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 — Verbatim Term: Neutropenic
Vomiting (Gastrointestinal disorders) | 2 — Verbatim Term: Emesis
Spleen Disorder (Blood and lymphatic system disorders) | 1 — Verbatim Term: Thrombocytopenia
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 — Verbatim Term: Glucose, uncontrolled
Paraesthesia (Nervous system disorders) | 2 — Verbatim Terms: Numbness of Hands, Numbness in Extremities
Dysuria (Renal and urinary disorders) | 1
Sleep Disturbance (Nervous system disorders) | 1
Hearing Impaired (Ear and labyrinth disorders) | 1 — Verbatim Term: Hearing Loss
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Bloating (Gastrointestinal disorders) | 1 — Verbatim Term: Burping
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 — Verbatim Terms: Left Upper Extremity (LUE) Pain; Left Lateral Thigh Pain
Pain (general) (General disorders) | 2 — Verbatim Terms: Left Upper Quadrant (LUQ) Pain; Right Upper Quadrant (RUQ) Pain
Blood in Stool (Gastrointestinal disorders) | 1
Thromboembolic Event (Vascular disorders) | 1 — Verbatim Terms: Deep Vein Thrombosis (DVT) in Right Lower Extremity; Superficial Vein Thrombosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03848182/Prot_SAP_001.pdf